CLINICAL TRIAL: NCT04311567
Title: Effects of Tofacitinib vs Methotrexate on Clinical and Molecular Disease Activity Markers in Joints and Lungs in Early Rheumatoid Arthritis (PULMORA) - A Randomized, Controlled, Open-label, Assessor-blinded, Phase IV Trial
Brief Title: Effects of Tofacitinib vs Methotrexate on Rheumatoid Arthritis Interstitial Lung Disease
Acronym: PULMORA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Low recruitment due to the pandemic and high screening failure rate in particular because of low prevalence of interstitial abnormalities at diagnosis in Sweden.
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EudraCT 2019-004179-38
Record Dates: First submitted 2020-03-05; First posted 2020-03-17 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2022-04

CONDITIONS: Rheumatoid Arthritis; Interstitial Lung Disease Due to Systemic Disease (Disorder); RA; ILD
Keywords: Rheumatoid arthritis; Interstitial lung disease; Janus Kinase inhibition; tofacitinib; methotrexate
MeSH Terms: conditions — Arthritis, Rheumatoid; Lung Diseases, Interstitial | interventions — tofacitinib; Methotrexate

STUDY DESIGN:
Intervention Model Description: A study in two parts:
  1. Screening with HRCT. Patients will be stratified based on the the findings to: cohort A, with pulmonary abnormalities; and cohort B, with normal findings (who will end further participation in the main trial).
  2. Randomization of cohort A to 48 weeks of active treatment. Parallel group design from baseline to week 24.
Who Masked: Outcomes Assessor
Masking Description: Blinded assessors of lung evaluation with HRCT and joint evaluation with joint counts (number of tender and swollen joints)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tofacitinib (Experimental): Oral tablet tofacitinib 5 mg BID for 48 weeks
  Interventions: Drug: Tofacitinib
- Methotrexate (Active Comparator): Oral tablet methotrexate 2.5 mg: 8 tablets in one dose (=20 mg) once weekly for 48 weeks
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Tofacitinib — Open-label tofacitinib for 48 weeks. All subjects (both arms) receive prednisone starting at 20 mg QD with tapering for 6 weeks. Patients with incomplete response at 24 weeks will escalate to combination therapy with tofacitinib 5 mg BID + methotrexate 20 mg weekly up to week 48.
  Other Names: Xeljanz
  Arms: Tofacitinib
Drug: Methotrexate — Open-label methotrexate for 48 weeks. All subjects (both arms) receive prednisone starting at 20 mg QD with tapering for 6 weeks. Patients with incomplete response at 24 weeks will escalate to combination therapy with tofacitinib 5 mg BID + methotrexate 20 mg weekly up to week 48.
  Other Names: metotrexat
  Arms: Methotrexate

SUMMARY:
Pulmonary abnormalities are present in up to 60% of patients with early rheumatoid arthritis (RA), and up to 10% of the patients will develop clinical interstitial lung disease (ILD). Recent data indicate that inhibition of Janus kinase is beneficial for this extra-articular manifestation. Our goal is to determine whether tofacitinib is an effective and safe treatment, compared to standard-of-care methotrexate, for subclinical and clinical ILD in patients with early RA. The study also explores disease mechanisms in lungs and joints, to identify potential biomarkers for diagnosis, prognosis, and response to treatment of RA-ILD.

DETAILED DESCRIPTION:
Study objectives:

Primary objective: Effects of tofacitinib compared to that of methotrexate on interstitial pulmonary abnormalities at 24 weeks.

Secondary objectives: Effects of tofacitinib compared to that of methotrexate on pulmonary abnormalities and function, RA disease activity and remission rates and patient reported outcome measures at different time points. Frequency of adverse events.

Exploratory objectives: Effects of tofacitinib compared to that of methotrexate on cellular and molecular activity profiles of clinical samples from joints and lungs.

Study design:

A randomized, actively controlled, open-label, assessor-blinded, multicenter 48 weeks phase IV trial. The study design includes an optional sub-study collecting tissue samples using ultrasound-guided synovial biopsies, bronchoalveolar lavage and Particles in Exhaled Air (PExA).

Study population and intervention:

Patients with early untreated RA with active and seropositive disease will be eligible for screening and the performance of high-resolution computed tomography (HRCT). Subjects with pulmonary abnormalities suggestive of RA-ILD will be randomized (1:1) to tofacitinib 5 mg BID (group 1) or standard-of-care methotrexate 20 mg weekly (group 2) for 48 weeks. All patients receive prednisone with tapering for 6 weeks. Patients with incomplete response at 24 weeks will escalate to combination therapy with tofacitinib+methotrexate (group 3). Intra-articular injections of cortisone will be allowed during the study.

145 subjects will be included and screened (part 1), and approximately 48 subjects will be randomized to active treatment (part 2).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of seropositive (i.e., presence of RF and/or anti-CCP antibodies) rheumatoid arthritis (RA) according to the ACR/EULAR 2010 criteria within 24 months.
2. No previous treatment with disease modifying anti-rheumatic drugs (DMARDs). History of prednisone use is allowed but should have been discontinued 2 weeks before baseline measurement.
3. Active disease with ≥2 painful and ≥2 swollen joints in 66/68 joints and CRP ≥2.0 mg/L
4. Aged 18-80 years
5. The subject has given written consent to participate in the study.

Exclusion Criteria:

1. Current active inflammatory joint disease other than RA.
2. Significant and/or uncontrolled cardiac, pulmonary disease, nervous system, renal, hepatic, endocrine or gastrointestinal disorders or severe RA which in the investigator's opinion would preclude patient participation.
3. Malignancy within the past 5 years, except for successfully treated cervical carcinoma in situ, basal cell and squamous cell carcinoma of the skin, with no evidence of recurrence or metastatic disease for at least 3 years.
4. Primary or secondary immunodeficiency (history of, or currently active), including known history of HIV infection.
5. Pregnant or lactating women.

   For subjects in part II the following exclusion criteria also apply:
6. Women of childbearing potential not willing or able to use highly effective methods of birth control per ICH M3 (R2) for 28 days prior and 3 months after end of study.
7. Active infection (excluding fungal infections of nail beds) requiring i.v. anti-infectives within 4 weeks, or oral anti-infectives within 2 weeks prior to baseline.
8. Positive tests for hepatitis B (HBsAg or HBV DNA),hepatitis C serology or SARS-CoV2
9. History of herpes zoster infection during last 10 years.
10. History or risk of venous thromboembolism or diverticulitis.
11. Positive tuberculosis history and/or positive Quantiferon test.
12. Hemoglobin <90 g/L.
13. Absolute neutrophil count < 1500 cells/uL.
14. ASAT or ALAT >2.0 times the upper limit of normal.
15. High or very high risk (≥ 5%) of cardiovascular death within 10 years by SCOREx1,5.
16. Multiple incidental solid/subsolid lung nodules of size ≥6 mm, single incidental solid lung nodules ≥8 mm.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-11-07 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-03-26 (Actual)

PRIMARY OUTCOMES:
Change in total interstitial disease score of pulmonary abnormalities by HRCT | Baseline and 24 weeks
  Total interstitial disease score will be calculated as the mean of six (anatomical levels) interstitial disease scores. Each level's interstitial disease score will be calculated as the sum of the extent of five different parenchymal patterns (Ground glass, reticulations, honey-combing, consolidations and emphysema) measured as percentage of pattern area to total lung area at a specified anatomical level.

SECONDARY OUTCOMES:
Change in extent of parenchymal lung disease by HRCT pattern | Baseline and 24 weeks
  The extent of the separate parenchymal pattern (Ground glass/reticulations/honey-combing/consolidations/emphysema) by HRCT measured as percentage of pattern area to total lung area at six different anatomical level.
Change in extent of parenchymal lung disease by HRCT pattern | Baseline and 48 weeks
  The extent of the separate parenchymal pattern (Ground glass/reticulations/honey-combing/consolidations/emphysema) by HRCT measured as percentage of pattern area to total lung area at six different anatomical level.
Change in Forced Vital Capacity (FVC) | Baseline and 24 weeks
  FVC will be measured by spirometry. The proportion of patients with FVC 24wks ≤ FVC baseline will also be calculated.
Change in Diffusion Capacity of Carbon Monoxide (DLCO) | Baseline and 24 weeks
  DLCO will be measured according to standard protocol and corrected for haemoglobulin level.
  Diffusion capacity divided by alveolar volume (DLCO/VA) will also be calculated.
Change in walking distance (meters) | Baseline and 24 weeks
  6-minutes walking test Diffusion capacity divided by alveolar volume (DLCO/VA) will also be calculated.
Change in blood oxygen saturation (SpO2) after 6-minutes walking | Baseline and 24 weeks
  6-minutes walking test with pulse oximetry recording Diffusion capacity divided by alveolar volume (DLCO/VA) will also be calculated.
Patient reported outcome of breathing and airway symptoms | baseline, 24 and 48 weeks
  Patient reported outcomes of breathing and airway symptoms will be evaluated using Saint George's Respiratory Questionnaire.
Disease activity score of rheumatoid arthritis (DAS28-CRP) | baseline, 12, 24 and 48 weeks
  DAS28-CRP will be calculated as follows: 0.56*√(TJC28) +0.28*√(SJC28)+0.014*PaGH+0.36*ln(CRP+1)+0.96.
  TJC = number of tender joints of 28, SJC= number of swollen joints of 28, CRP=c-reactive protein level and PaGH=Patient reported global impact of disease on health on a VAS scale (0-100)
Patient reported health assessment of physical function (HAQ index) | baseline, 24 and 48 weeks
  Patient reported function assessed by a validated questionnaire HAQ = health assessment questionnaire. The assessment gives a value/index between 0 - 3.0.
Proportion of patients in rheumatoid arthritis DAS remission | 24 and 48 weeks
  DAS28 remission is defined as DAS28<2.6.
Frequency of adverse events (AE) | baseline, 24 and 48 weeks
  Number of AE per category and serious AE will be calculated for the different treatment groups
Patient reported global disease activity | baseline, 12, 24 and 48 weeks
  Patient reported global impact of disease on health on a VAS scale (0-100 mm)
Proportion of patients in rheumatoid arthritis ACR-EULAR Boolean remission | 24 and 48 weeks
  Boolean RA remission is defined as: SJC, TJC, PaGH and CRP, all ≤1. TJC = number of tender joints of 28, SJC= number of swollen joints of 28 and PaGH=Patient reported global impact of disease on health on a VAS scale (0-10)
Clinical disease activity score of rheumatoid arthritis (CDAI) | baseline, 12, 24 and 48 weeks
  Clinical disease activity score of rheumatoid arthritis (CDAI) is calculated as follows: SJC + TJC + PaGH + PhGH.
  TJC = number of tender joints of 28, SJC= number of swollen joints of 28, PaGH=Patient reported global impact of disease on health on a VAS scale (0-10) and PhGH=physician assessment of global impact of disease on health of patient on a VAS scale (0-10). CDAI ranges from 0 - 76.

OTHER OUTCOMES:
Change in cellular activity profile of clinical samples | baseline and 24 weeks
  Exploratory sub-study: Frequencies (% of total cell populations) of subtypes of immune- and stroma cells (defined by a core set of cell surface markers) isolated from synovial biopsies and broncho-alveolar lavage samples and evaluated by flowcytometry
Change in molecular activity profile of clinical samples | Baseline and 24 weeks
  Exploratory sub-study: Gene expression of bulk tissue and sorted cells of synovial biopsies and broncho-alveolar lavage samples by RNA sequencing. Levels of cytokines (IL-1β, IFN-α2, IFN-γ, TNF-α, IL-6, IL-8 (CXCL8), IL-10, IL-12p70, IL-17A, IL-18, IL-23, and IL-33), chemokines (CCL2, CCL3, CCL4, CCL5, CCL11, CCL17, CCL20, CXCL1, CXCL5, CXCL8, CXCL9, CXCL10, CXCL11) and growth factors (GM-CSF, PDGF and TGFbeta1) of synovial fluid, blood and broncho-alveolar lavage will be determined by bead-based immunoassay.
  Clinical fluid droplet samples containing lipids and proteins from small airways will be collected on a membrane using a novel non-invasive method - Particles in Exhaled Air (PExA) and analyzed using mass spectrometry.

CONTACTS AND LOCATIONS:
Overall Officials: Anna-Karin H Ekwall, MD MSc PhD, Principal Investigator — The Sahlgrenska University Hospital and University of Gothenburg
Locations (3):
- Sweden (3):
  - Skåne University Hospital, Department of Rheumatology, Lund, Skåne County
  - Clinical Rheumatology Research Center, The Sahlgrenska University Hospital, Gothenburg, Västra Götaland County
  - Karolinska University Hospital, Department of Rheumatology, Stockholm